CLINICAL TRIAL: NCT02194010
Title: Disability Severity Scale (DSI) and Hereditary Motor and Sensory Neuropathy Overall Disability Scale (HMSN-R-ODS)
Acronym: DSI and HMSN
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Charcot-Marie-Tooth Association (Other); Muscular Dystrophy Association (Other); University of Rochester (Other); University of South Florida (Other)
Responsible Party: Principal Investigator, Michael Shy, Professor of Neurology, University of Iowa
Other Study IDs: INC 6610; U54NS065712 (NIH)
Record Dates: First submitted 2014-04-02; First posted 2014-07-18 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Charcot Marie Tooth Disease; Inherited Peripheral Neuropathy
Keywords: Outcome Measure; Patient Reported Questionnaires
MeSH Terms: conditions — Charcot-Marie-Tooth Disease; Inherited Peripheral Neuropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Participants evaluated at INC sites: Participants being evaluated at the INC sites will participate in both the DSI and HMSN-R-ODS by completing these PROs during their visit.
- INC Contact Registry: INC Contact Registry completes the HMSN-R-ODS on web http://rarediseasesnetwork.epi.usf.edu/INC/

SUMMARY:
The purpose of this research study is to create and validate two patient reported outcome (PRO) questionnaires. PRO questionnaires ask questions that help to measure disability in patients with inherited neuropathies. These questionnaires ask questions about what participants think disability is for themselves or others with inherited neuropathies. These questionnaires are a useful tool when evaluating whether treatments are working in the day to day life of an individual, although there are currently no questionnaires available specifically for people who have Charcot Marie Tooth disease (CMT).

DETAILED DESCRIPTION:
Charcot Marie Tooth Disease (CMT) is a group of disorders that cause a peripheral neuropathy, impairing the long nerves that go to the feet and hands. Due to the problems with the peripheral nerves, people with CMT have muscle weakness and sensory loss that impairs their physical abilities. CMT affects approximately 1 in 2500 people and is caused my mutations in over 70 different genes. Models exist for many sub-types of CMT that have led to an increased understanding of the biological basis for these disorders. These advances have also made rational therapies for CMT a realistic possibility. However, clinical trials have been limited in CMT by a combination of lack of natural history data for many subtypes, a lack of outcome measures that can detect change in a short period for slowly progressive forms of CMT, and a lack of outcome measures for young children with CMT.

In order to develop treatments based on the biological advances in the inherited neuropathies, it is necessary to have measured the natural history of the various disorders. It is only by knowing the natural history that one understands the onset of clinical symptoms, the rate of progression, and the ultimate prognosis of these diseases. For these reasons, the INC has dedicated much of its effort to develop sensitive outcome instruments, including PRO tools, to measure the natural history of CMT. It is the investigators goal to establish such an instrument for overall impairment for use in both natural history analysis and clinical trials. To develop and validate this instrument, the investigators will be asking people who have CMT to complete two questionnaires, the DSI and the HMSN-R-ODS. These relate to overall symptom impairment due to CMT. These instruments may be used to help us understand the overall progression of CMT and will ultimately help with clinical trials when they are available for the various forms of CMT.

ELIGIBILITY:
Inclusion Criteria:

* individual has an inherited peripheral neuropathy or is suspected to have an inherited peripheral neuropathy
* individual is 10-99 years of age
* individual signs consent or assent form depending on age and requirements
* individual is participating in INC 6601 at one of the participating sites OR is a participant on the INC Patient Registry

Exclusion Criteria:

* inability to provide informed consent
* outside of age range
* inability to complete questionnaire
* does not understand English
* is not participating in INC 6601 or on the INC Patient Registry

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants enrolled in INC protocol 6601 and being seen at a participating site for an evaluation of CMT will be asked if they would like to participate in this protocol. The individuals being recruited will have already signed consent forms and be enrolled in 6601. They will be informed that it is completely voluntary to participate in this protocol, and they can still be enrolled in INC 6601 without participating in this project.
  Alternative participants who are registered with our INC Patient Registry will be alerted to the form through an email and asked to participate due to their diagnosis of suspected diagnosis of CMT.
Sampling Method: Non-Probability Sample
Enrollment: 563 (Actual)
Dates: Start 2014-04; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Disability Severity Index | Approximately 30 minutes
  The DSI asks the subject to provide information about how disability is reflected in general by equipment required for mobility. Therefore, the DSI asks the subject if a person in general was wearing AFOs (braces) for mobility, what level of disability would that reflect using both a quantitative measurement of score and a verbal method of scoring (none, mild, moderate, severe). These questions do not apply to the participant themselves, just in general how disabled they believe a person to be based on the mobility assistive devices that that person requires. Then a research team member will complete the last page which specifically asks about what that subject is using for mobility.

SECONDARY OUTCOMES:
Hereditary Motor and Sensory Neuropathy Overall Disability Scale (HMSN-R-ODS) | Approximately 30 minutes
  The HMSN-R-ODS is a functional score about the subject asking about their daily activities and overall health. Questions are grouped in various sections and include: Changing and holding body positions; walking and movement; movement by transport; carrying, moving, or handling objects; self-care; household activities and duties; taking care (daily tasks) - general; meeting other people; work, study, and hobbies. These questions relate specifically to the subject and ask how they can perform these various activities with little to severe difficulty.

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Shy, MD, Principal Investigator — Universit of Iowa
Locations (3):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - University of Rochester Medical Center, Rochester, New York
- National Hospital of Neurology and Neurosurgery, London, United Kingdom